CLINICAL TRIAL: NCT03524482
Title: Development and Pilot Evaluation of the Path2Quit Tobacco Intervention Targeting African Americans
Brief Title: Path2Quit Tobacco Intervention For African Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CASE1Y18
Record Dates: First submitted 2018-04-30; First posted 2018-05-14 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Smoking Cessation; Smoking, Tobacco
Keywords: culturally specific
MeSH Terms: conditions — Smoking Cessation; Tobacco Smoking

STUDY DESIGN:
Intervention Model Description: We will conduct a 2-arm semi-pragmatic randomized design among current tobacco users (N=100). CMHA residents will be randomly assigned to receive (1) the newly translated Path2Quit or (2) SmokeFreeText (NCI's publicly available, standard text messaging program) combined with brief behavioral counseling session plus 2 weeks of nicotine replacement therapy (NRT).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Path2Quit (Experimental): Culturally specific text message intervention
  Interventions: Behavioral: Path2Quit
- SmokeFreeText (Active Comparator): The National Cancer Institute's publicly available, standard text messaging program for tobacco cessation
  Interventions: Behavioral: SmokeFreeText

INTERVENTIONS:
Behavioral: SmokeFreeText — SmokefreeTXT is a 6-8 week fully automated text-based cessation intervention. The program is free to U.S. subscribers who have a mobile phone, and is available on smokefree.gov or by texting "QUIT" to short code 47848. Participants are encouraged to set a quit date within the next 14 days, followed by count-down messages leading to the quit date. Starting on the quit date, participants receive 6 weeks of intervention text messages, and assessment questions (mood, cravings, smoking status). The message library contains 166 messages and 41 behavior change techniques,40 which are delivered at the greatest frequency during the first 2 weeks and taper over time. When in need of assistance, participants can text one of 3 keywords (MOOD, CRAVE, or SLIP) to receive a relevant message from the system. Participants can opt-out by texting STOP at any time. With informed consent, we will be able to access the SmokefreeTXT data for these participants.
  Other Names: SmokefreeTXT
  Arms: SmokeFreeText
Behavioral: Path2Quit — Path2Quit will deliver 20-60 second video clips by multimedia messaging service. The message library will include 75-170 messages. Written text messages will be limited to brief phrases to indicate the topic of the video. Messages will be pushed to participants in the morning, in the afternoon, and 2 hours before the reported usual bedtime. The cultural adaptations will be infused throughout the video segments. Topics include deep structure: race and smoking in general, African American smoking statistics; norms for smoking; concerns about nicotine replacement/medication; family/collectivism; unique stressors; racism/discrimination, depression; co-morbid addiction; neighborhood/environmental influences; menthol cigarettes; race-specific weight issues and concerns; and working as a community against the tobacco industry.
  Arms: Path2Quit

SUMMARY:
The purpose of this research is to study a smoking cessation program for adult smokers in Northeast Ohio. The study will also look at how different people respond to the program.

The study includes completing surveys and receiving text messages to help participants become tobacco free.

DETAILED DESCRIPTION:
OBJECTIVES Specific Aim 1: Translate a culturally specific video-based tobacco use intervention into a scalable mobile health (mhealth) format.

Specific Aim 2: Conduct a pilot study of the video-text intervention.

Study Design:

2-arm semi-pragmatic randomized design among current tobacco users

Cuyahoga Metropolitan Housing Authority residents will be randomly assigned to receive (1) the newly translated Path2Quit or (2) SmokeFreeText (NCI's publicly available, standard text messaging program) combined with brief behavioral counseling session plus 2 weeks of nicotine replacement therapy (NRT). Primary outcomes will include intervention evaluations (content and format), acceptability, coping strategies, engagement, and NRT adherence. Secondary variables will include 24-hour quit attempts and biochemically verified tobacco use abstinence at the 1-month follow-up. Exploratory mediational analyses will examine the roles of urban hassles, acculturation, neighborhood environment, ethnic discrimination, and psychological distress in intervention effects.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as African American
* Either smoke at least 1 cigarettes/day or have a carbon monoxide (CO) reading of at least 4 ppm
* Consistent with SmokefreeTXT, be willing to set a quit date within the next 14 days.
* Recruited from Cleveland metropolitan housing authority or who report low income based on federal guidelines

Exclusion Criteria:

* Does not meet all of the above inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-08-20 (Actual); Study Completion 2018-08-20 (Actual)

PRIMARY OUTCOMES:
Proportion of participants who abstain from smoking | At 1-month follow-up
  Abstinence will be coded as a binary variable. Analysis will be conducted with an intent to treat approach

SECONDARY OUTCOMES:
Number of missed nicotine replacement therapy doses | Up to 1-month follow-up
  Measure of NRT adherence. Number of missed doses will be recorded for each participant
24-Hour quit attempts | At 1-month follow-up
  Number of times a participant quits smoking for at least 24 hours
Changes in carbon monoxide breath levels from baseline to followup | At 1-month follow-up
  Breath carbon monoxide tests will biochemically confirm self-reported cessation
Changes in Contemplation ladder score | From baseline to up to 1-month follow-up
  self-reported score 0-10 where a higher score indicates more readiness to quit
Average score of Intervention Evaluation (IRQ) | At 1-month follow-up
  The IRQ is a 22 item scale scored 0-7 (total score 0-154) where higher scores indicate more satisfaction
Average score of smoking urges | Up to 1-month follow-up
  This brief, 10 item scale is scores 1-7 (total score 10-70) with higher scores indicating greater agreement

OTHER OUTCOMES:
Average scores of Urban hassles | Changes from baseline to 1 month follow-up
  This is a 63 item scale scored 0-5 (total score 0-315) where higher scores indicate more severe hassle
Average Neighborhood Environment scale score | At Baseline
  The neighborhood environment scale is an 18 item True or False scale
Average General Ethnic Discrimination Scale Score | At baseline
  This is a measure of ethnic discrimination. These 16 items are scored 1-6 (total score 16-96) with higher scores indicating greater levels of ethnic discrimination
Average psychological distress score using the the perceived stress scale | At baseline
  A ten item scale with each item scored 0-4 (total score 0-40) where higher scores indicate more stress. Positive items are scored in reverse.
Average depression score using Center for Epidemiological Studies Depression (CES-D) Scale | At baseline
  A twenty item scale ranging from 0-60 with each item scored 0-3. Higher scores indicate more depression
Average Beliefs and Attitudes Survey Score | At baseline
  This is a 24 item scale (total range 24-168) with each item scored 1-7. Higher scores indicate greater levels of agreement
Average Ethnic Identity Score | At baseline
  This is based on the Multigroup Ethnic Identity Measure scale. These five items are scored 1-4 for a total score of 5-20. Higher scores indicate stronger ethnic identity
Average Culturally Specific Interventions Expectancy Questionnaire | At baseline
  The Culturally Specific Interventions Expectancy Questionnaire is a 2 item scale with each item ranging 1-5 (total score 2-10) where higher scores indicate greater agreement.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Webb Hooper, PhD, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- Case Western Reserve University, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Webb Hooper M, Miller DB, Saldivar E, Mitchell C, Johnson L, Burns M, Huang MC. Randomized controlled trial testing a video-text tobacco cessation intervention among economically disadvantaged African American adults. Psychol Addict Behav. 2021 Nov;35(7):769-777. doi: 10.1037/adb0000691. Epub 2021 Oct 14. PMID 34647777